CLINICAL TRIAL: NCT05870228
Title: Investigating the Feasibility, Acceptability, and Preliminary Effectiveness of a Sleep Intervention for Adolescents With Co-morbid Insomnia and Mental Health Difficulties
Brief Title: Investigating a Sleep Intervention for Adolescents Attending Mental Health Services
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was 'completed' within allocated timeframe. However, we were unable to recruit the initial target number of adolescent participants, thus concluding it is not currently feasible to recruit adolescents to complete the intervention.
Sponsor: Stephanie McCrory (Other)
Responsible Party: Sponsor-Investigator, Stephanie McCrory, Principal Investigator, University of Strathclyde
Organization: University of Strathclyde (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UEC2331
Record Dates: First submitted 2023-04-24; First posted 2023-05-23 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Insomnia; Mental Health Issue
Keywords: Adolescent Sleep; Insomnia; Mental Health; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm intervention group (Other): Single-arm intervention
  Interventions: Behavioral: Strathclyde Sleep Intervention

INTERVENTIONS:
Behavioral: Strathclyde Sleep Intervention — Manual-based CBT-I

SUMMARY:
The overall objectives of the study are to:

1. To assess the feasibility of delivering the Strathclyde Sleep Intervention to adolescents with co-morbid insomnia and mental health attending a mental health services The following feasibility benchmarks will be assessed: recruitment and retention, participant attendance, staff training, intervention fidelity and participant adherence.
2. To examine participant acceptability. The researchers will conduct qualitative interviews with the participants and delivery staff to examine the acceptability of the programme.
3. To investigate the preliminary effectiveness by assessing the following: sleep parameters, insomnia symptoms, Circadian phase preference (baseline only) and mental health symptoms. Data will be collected at baseline, post-intervention and 3 month follow-up.

DETAILED DESCRIPTION:
Sleep problems have a significant detrimental impact on physical health, development, and functioning and are commonly experienced co-morbidly with other mental health problems. Therefore, many adolescents who are attending mental health services, also experience significant sleep disturbances. However, sleep problems are rarely addressed within mental health services due to lack of awareness of the importance of sleep and/or training in effective treatments. Cognitive behavioural therapy for insomnia (CBT-I) is the recommended approach for treating insomnia in both adult and adolescent populations. Despite this, there has been limited research investigating the delivery of CBT-I interventions to adolescents with co-morbid mental health problems, and to our knowledge, no such studies exist within the Scottish context. The Strathclyde Sleep Intervention incorporates CBT-I components to improve adolescent sleep. This study aims to evaluate the feasibility, acceptability, and preliminary effectiveness of the intervention for adolescents attending mental health services. Staff within the service will receive training to deliver the Strathclyde Sleep Intervention to adolescents with co-morbid mental health and sleep problems. The following feasibility benchmarks will be assessed: recruitment and retention, participant attendance, facilitator training, intervention fidelity and participant adherence. Acceptability will be measured via qualitative interviews with participants and staff. Baseline, post-intervention, and follow-up assessments will be conducted to assess preliminary effectiveness of the intervention for improving sleep and mental health. This research is necessary to inform future trials of the Strathclyde Sleep Intervention and to support its wider implementation within services.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents (12-15 years)
2. Meeting thresholds for insomnia disorder (determined by cut-off scores on the 2 item Sleep Condition Indicator (score <2 indicates probable insomnia)
3. Attending CAMHS for mental health intervention/support
4. Able to engage with intervention protocol

Exclusion Criteria:

1. Active suicide ideation and/or recent suicidal attempts
2. Contraindicators for components of CBT-I (sleep restriction therapy) including seizure disorders/conditions including epilepsy, bipolar disorder, symptoms of psychosis, obstructive sleep apnea and parasomnias.
3. Diagnosis of Autism Spectrum Disorder, Attention Deficit Hyperactivity Disorder, Foetal Alcohol Spectrum Disorder (Neurodiversity)
4. Those who are currently completing, or have recently completed (in the past 6 months), CBT-I for insomnia elsewhere (or components of CBT-I including e.g. sleep restriction therapy, stimulus control, cognitive techniques). This will only include in-person, one-to-one methods of delivery

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Fleming, PhD, Principal Investigator — University of Strathclyde
Locations (1):
- East Renfrewshire Healthier Minds Team, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from 2 mental health services in Scotland
Groups:
- Adolescent Participants: Single-arm intervention comprised of adolescent participants
  Strathclyde Sleep Intervention: Manual-based CBT-I
- Practitioner Participants: Practitioner participants recruited to complete training, deliver the intervention and/or participate in interview.
Period: Overall Study
Arm/Group | Adolescent Participants | Practitioner Participants
Started | 3 | 13
Completed | 0 (1 participant completed 1/4 sessions, 1 participant completed 3/4 sessions, 1 participant completed 4/4 sessions. No participants completed the post-intervention or follow-up assessment(s) and/or qualitative feedback.) | 13
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: 3 adolescent participants
  13 practitioner participants
Groups:
- Adolescent Participants: Single-arm intervention comprised of adolescent participants (n=3)
- Practitioner Participants: Practitioner participants recruited to complete training, deliver the intervention and/or participate in interview (n=13)
- Total: Total of all reporting groups
Arm/Group | Adolescent Participants | Practitioner Participants | Total
Number analyzed (Participants) | 3 | 13 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 0 | 13 | 13
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: There was low numbers of adolescents recruited (n = 3), poor retention rates (2 lost to follow-up, & 1 withdrew) and lack of post-intervention or follow-up data. No adolescents participated in the qualitative interviews. Therefore, there was 13 practitioner participants who completed the qualitative interviews.
  years | 15.33 (1.24) | 38 (10) | 33.69 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: There was low numbers of adolescents recruited (n = 3), poor retention rates (2 lost to follow-up, & 1 withdrew) and lack of post-intervention or follow-up data. No adolescents participated in the qualitative interviews. Therefore, there was 13 practitioner participants who completed the qualitative interviews.
  Participants
    Female | 2 | 12 | 14
    Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 3 | 13 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Adolescent Participants Recruited
Description: A total of 8 adolescents were referred between October 2023 and October 2024. Of these, 1 was ineligible, 4 declined participation / did not respond, and 3 provided consent and were enrolled.
Time Frame: 1 year
Population: Adolescents referred to the study (N = 7 eligible participants)
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent Participants: Adolescent participants who consented to participate in the intervention feasibility study.
Arm/Group | Adolescent Participants
Number analyzed (Participants) | 7
Participants | 3

2. Primary Outcome: Number of Adolescent Participants Who Attend Each Session
Description: Measured through attendance logs. This outcome reports the number of adolescent participants who completed each session of the 4-session intervention.
Time Frame: Over 4 session intervention period (1 - 4 months) 1-4 months 1-4 months
Population: Adolescents
Measure: Count of Participants; unit: Participants
Groups:
- Adolescent Participants: Adolescent participants who received the Strathclyde Sleep Intervention (manual-based CBT-I) as part of the feasibility study.
Arm/Group | Adolescent Participants
Number analyzed (Participants) | 3
Participants
  Completed all sessions | 1
  Completed 3 sessions | 1
  Completed 1 session | 1

3. Primary Outcome: Intervention Fidelity
Description: Fidelity was assessed using an intervention delivery checklist. Practitioners were categorised based on whether they delivered the intervention as intended or deviated. Of the 10 practitioners who completed training, only 3 practitioners delivered the intervention, but only 2 submitted fidelity data for this outcome.
Time Frame: 1-4 months
Population: Practitioners who delivered the intervention and submitted recordings for fidelity assessment.
Measure: Number; unit: participants
Groups:
- Practitioner Participants: Practitioner participants only. Of the 3 practitioners who delivered the intervention, only 2 submitted session recordings. A total of 5 sessions were recorded and reviewed for fidelity.
Arm/Group | Practitioner Participants
Number analyzed (Participants) | 2
participants
  Delivered intervention as intended | 2
  Deviated from intended delivery | 0

4. Secondary Outcome: Acceptability of Intervention to Practitioners
Description: Measured through qualitative interviews conducted with mental health practitioners and service managers (N = 13) to explore their experiences of the intervention and feasibility of delivery in practice.
Time Frame: Up to 9 months post-training
Population: Mental health practitioners who received training and service managers who overseen the implementation of the intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Practitioner Participants: Practitioner participants
Arm/Group | Practitioner Participants
Number analyzed (Participants) | 13
Participants
  Sleep problems are common, but they are poorly assessed and treated | 13
  The training and CBTi intervention was acceptable for practitioners in mental health services | 13
  The CBTi intervention may not be suitable for most adolescents attending mental health services | 12
  CBTi must be delivered flexibly, balancing patient need and available resource | 13
  'Red tape' restrictions make conducting research in mental health services challenging | 12

5. Secondary Outcome: Sleep Outcomes (Change From Baseline, Post-intervention and Follow-up)
Description: Sleep outcomes were intended to be assessed using a consensus sleep diary completed by adolescent participants at three time points: baseline (2 weeks prior to intervention), post-intervention (2 weeks after intervention), and follow-up (3 months after intervention).
  However, only baseline data were completed by 3 participants. No post-intervention or follow-up sleep diary data were collected.
  This table summarizes baseline sleep outcomes only, based on the sleep efficiency score - a key sleep parameter calculated as:
  Sleep Efficiency (%) = (Total Sleep Time / Time in Bed) × 100
  Higher scores indicate better sleep efficiency, with scores above 90% typically considered good.
Time Frame: Baseline (2 weeks before intervention delivery)
Population: All 3 adolescent participants completed baseline sleep assessments. No participants completed post-intervention or follow-up assessments.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adolescent Participants: Single arm Adolescent participants
Arm/Group | Adolescent Participants
Number analyzed (Participants) | 3
units on a scale | 84.71 (11.64)

6. Secondary Outcome: Insomnia Symptoms Assessed Using Sleep Condition Indicator (Score of <16 Indicates Probable Insomnia, Higher Scores Indicate Better Sleep, Scores Range 0-32) (Change From Baseline, Post-intervention and Follow-up)
Description: Insomnia symptoms were intended to be measured using the Sleep Condition Indicator (SCI), completed by adolescent participants at three time points: Baseline (2 weeks prior to intervention), Post-intervention (2 weeks following intervention), Follow-up (3 months post-intervention)
  Sleep Condition Indicator scores range from 0-32, with higher scores indicating better sleep. A score <16 suggests probable insomnia. However, only baseline SCI scores were collected from participants. No post-intervention or follow-up data were submitted.
Time Frame: Baseline (2 weeks before intervention) Baseline (2 weeks before intervention) Baseline (2 weeks before intervention)
Population: Adolescents - Baseline only as none completed post-intervention or follow-up outcome measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adolescent Participants: Single arm - Adolescent participants only
Arm/Group | Adolescent Participants
Number analyzed (Participants) | 3
score on a scale | 7 (1)

7. Secondary Outcome: Depression and Anxiety Symptoms Assessed by Revised Child Anxiety and Depression Scale - 25 Item Version (RCADS-25) (Change From Baseline, Post-intervention and Follow-up)
Description: Symptoms of depression and anxiety were intended to be assessed using the Revised Child Anxiety and Depression Scale - 25 item version (RCADS-25), completed by adolescent participants at three time points: Baseline (2 weeks prior to intervention), Post-intervention (2 weeks after intervention), Follow-up (3 months after intervention)
  RCADS-25 provides total scores and subscale scores for anxiety and depression. The anxiety subscale includes 15 items and scores range from 0-45. The depression subscale comprises 10 items and scores range from 0-30. A total score can be calculated by summing the depression and anxiety subscales and the total scores range from 0-75. Higher scores on any subscale or the total score represent greater symptom severity.
  However, only baseline data were collected. No post-intervention or follow-up RCADS-25 data were submitted by any of the 3 adolescent participants
Time Frame: Baseline (2-weeks before intervention delivery)
Population: Baseline RCADS-25 scores were submitted by 3 adolescent participants. No post-intervention or follow-up data were collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescent Participants
Number analyzed (Participants) | 3
score on a scale
  Depression sub-scale | 14 (7.94)
  Anxiety subscale | 17.67 (5.69)
  Total score | 31.67 (13.65)

8. Secondary Outcome: Anxiety Symptoms Measured by GAD-7 (Change From Baseline, Post-intervention and Follow-up)
Description: Measured by Generalised Anxiety Disorder Assessment (GAD-7). The GAD-7 will be utilised to measure symptoms of anxiety. The measure consists of 7 items assessing anxiety symptoms over the previous 2 weeks. Scores range from 0-21, higher scores indicate greater symptom severity (5- mild, 10 - moderate, 15- severe). We intended to collect data at three time points: Baseline (2 weeks prior to intervention), Post-intervention (2 weeks after intervention), Follow-up (3 months after intervention)
  However, only 1 participant completed this measure at baseline. No post-intervention or follow-up GAD-7 data were submitted by participants.
Time Frame: Baseline (2-weeks before intervention delivery)
Population: Baseline GAD-7 scores were submitted by 3 adolescent participants. No post-intervention or follow-up data were collected.
Measure: Number; unit: score on a scale
Arm/Group | Adolescent Participants
Number analyzed (Participants) | 1
score on a scale | 11

9. Secondary Outcome: Depression Symptoms Measured by PHQ-9 (Change From Baseline, Post-intervention and Follow-up)
Description: Depression symptoms were intended to be measured using the Patient Health Questionnaire-9 (PHQ-9) at three time points:
  Baseline (2 weeks prior to intervention), Post-intervention (2 weeks after intervention), Follow-up (3 months after intervention)
  The PHQ-9 consists of 9 items, each scored 0-3, with total scores ranging from 0-27. Higher scores indicate more severe depressive symptoms. However, only baseline PHQ-9 data were submitted by participants. No post-intervention or follow-up data were collected.
Time Frame: Baseline (2-weeks before intervention delivery)
Population: Adolescents - Baseline only. None completed post-intervention or follow-up assesments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescent Participants
Number analyzed (Participants) | 3
score on a scale | 15.33 (7.51)

10. Secondary Outcome: Circadian Phase Preference Measured by Morningness/Eveningness Scale for Children
Description: Measured by Morningness/eveningness scale for children (MESC). This 10-item measure will be used to assess circadian phase preference. Items are scored on from 1- 5 item scale and scores range from 10-42. Lower scores indicate greater eveningness (<20) and higher scores indicate greater morningness (>28). This item will be collected in the baseline assessment.
Time Frame: Baseline only
Population: Adolescents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescent Participants
Number analyzed (Participants) | 3
score on a scale | 21.33 (2.89)

11. Other Pre Specified Outcome: Staff Satisfaction With Training
Description: Satisfaction with the training was assessed through qualitative interviews with practitioner participants. This outcome includes only those who completed the training (10 out of 13 participants).
Time Frame: Up to 9 months post-training
Population: All practitioners who completed training (n=10)
Measure: Count of Participants; unit: Participants
Groups:
- Practitioner Participants: Practitioners who received and completed the training.
Arm/Group | Practitioner Participants
Number analyzed (Participants) | 10
Participants
  Staff were satisfied with training | 10
  Staff not satisfied with training | 0

ADVERSE EVENTS:
Time Frame: up to 6 months
Description: Adverse events will be monitored throughout the intervention and will be defined as either unrelated, possibly unrelated, probably, or definitely related to the intervention. Serious adverse events will be defined as reactions that threaten life or functioning. In line with the CONSORT guidelines, adverse events will be defined as anticipated or unexpected. Deaths and Adverse Events not assessed for practitioners.
Arm/Group | Adolescent Participants
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adolescent Participants (N=3)
Social circumstance, unexpected & possibly related (Social circumstances) | 1 (1) — Participant experienced a deterioration in mental health while participating. The event was deemed as unexpected, possibly related. The participant decided to withdraw and appropriate support was in place via mental health practitioner.

LIMITATIONS AND CAVEATS:
Recruitment and retention of adolescents was challenging. Key barriers included: most adolescents had diagnosis of NDD (exclusion criteria), time pressure and demands on the services made it difficult to implement. Qualitative feedback only obtained from practitioners, therefore, not able to examine acceptability from adolescents' perspective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT05870228/Prot_SAP_000.pdf